CLINICAL TRIAL: NCT06108076
Title: Acute and Chronic Effects of Oral Ketones in Subjects With HFrEF and Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230420HU; 1UM1TR004538-01 (NIH)
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Heart Failure, Reduced Ejection Fraction
Keywords: Ketone esters; Cardiopulmonary benefits; Left Ventricular function; Stroke volume; Cardiac output
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure, Systolic | interventions — rVSV-deltaG-spike COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Open label, pilot trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketone Ester administration (Experimental): 1. Monitored administration of oral Ketone monoester at 400mg/kg dosed twice on visit 2 (cardiac MRI day)
  2. Self administered oral β-hydroxybutyrate (BOHB) at 400mg/kg/day for a period of 6 days
  Interventions: Drug: Ketone Monoester (KE)

INTERVENTIONS:
Drug: Ketone Monoester (KE) — Ketones are a nutritional supplement currently used by athletes for their performance enhancing effects - specifically their cardio-pulmonary benefits
  Other Names: DeltaG

SUMMARY:
This study will provide insight into whether cardiac function changes with oral Ketone Esters (KE) administered to patients with Type 2 Diabetes Mellitus (T2DM) and Heart failure with reduced ejection fraction (HFrEF). Plasma ketones are avidly extracted by cardiac muscle and their uptake is not dependent upon insulin or influenced by insulin resistance.

DETAILED DESCRIPTION:
After the screening visit, subject will take two separate doses of oral ketones during visit two. Subjects will have their first dose (400mg/kg) upon completion of the baseline Magnetic Resonance Imaging (MRI), and then a second dose (400mg/kg) approximately 1.5 hours after their consumption of the 1st dose. Approximately 1.5 hours after their second dose (3hr since first dose), the subject will undergo a second cardiac MRI. Baseline Blood samples of Beta-hydroxybutyrate (BOHB), acetoacetate (ACAC), Free Fatty Acids (FFA), insulin, c-peptide, glucagon, and an additional 10ml (for storage and later analysis) will be drawn prior to their first dose, then every 30 minutes after their first dose, until completion of the second MRI, then a final blood draw upon completion of the MRI for a total of 8 blood draws during visit 2. An IV catheter will be placed into one antecubital vein by a study nurse for all blood draws during visit 2.

The subject will then be asked to return to complete a third MRI approximately 24 hours after their second MRI. Blood samples for BOHB, acetoacetate (ACAC), insulin, c-peptide and glucagon, and an additional 10 ml will be drawn prior to their third MRI. An IV catheter will be placed into one antecubital vein by a study nurse for all blood draws during visit 3.

After completion of the third MRI, subjects will be dosed KE 400mg/kg once daily until the visit 4 MRI can be completed.

Blood samples for BOHB, acetoacetate (ACAC), insulin, c-peptide, glucagon, proBNP, and an additional 10 ml will be drawn prior to their fourth MRI. An IV catheter will be placed into one antecubital vein by a study nurse for all blood draws during visit 4. The 4th MRI, based on subject and scanner availability at approximately Day 7

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be on a stable dose of guideline-directed medications for Heart Failure (HF).
* Patients will have an established diagnosis of HF before the screening visit, documented by an acceptable imaging modality in the last 6 months.
* Age = 18-80 y
* Body Mass Index (BMI) =23-38 kg/m2
* Glycated hemoglobin (HbA1c) = 6.0-10.0%
* Blood Pressure (BP) < 145/85 mmHg
* Estimated Glomerular Filtration Rate (eGFR) > 30 ml/min•1.73 m2
* For women of child-bearing age (WOCBA) willingness to use contraception, if applicable.

Exclusion Criteria:

* Patients treated with Sodium-Glucose Transport Protein (SGLT2i's) or medications that may impair heart function or acutely worsen glycemic control will be excluded.
* Pregnancy, lactation, or plans to become pregnant. A negative pregnancy test will be performed before each Magnetic resonance imaging (MRI) study to assess current status.
* Allergy/sensitivity to study drugs or their ingredients.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Subjects with a history of cancer (except basal or squamous cell cancer that has been resolved/remission for 5 years)
* Cardiovascular event within the last 3 months
* Major organ or metabolic diseases, or physical limitations that will not allow the subject to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Efficiency after acute dose (Left-ventricular function) | 1.5 hours to 24 hours
  Change in cardiac efficiency after acute dosing of KE, measured by change in Left-ventricular function measured using Cardiac MRI and expressed as a percentage.
Cardiac Efficiency after chronic dosing (Left-ventricular function) | 1.5 hours to 7 days
  Change in cardiac efficiency after chronic (7 day) dosing of KE, measured by change in Left-Ventricular function measured using Cardiac MRI and expressed as a percentage.

SECONDARY OUTCOMES:
Six minute walk test | Baseline to 7 days
  Participants will be asked to walk as far as possible for 6 minutes, escorted by a member of the research team.
  Baseline to 7 day distance will be compared.
Acetoacetate | Baseline to 7 days
  Baseline to 7 day level will be compared.
Glucose | Baseline to 7 days
  Baseline to 7 day level will be compared.
Free Fatty Acids (FFAs) | Baseline to 7 days
  Baseline to 7 day level will be compared.
Insulin/C-peptide | Baseline to 7 days
  Baseline to 7 day level will be compared.
Glucagon | Baseline to 7 days
  Baseline to 7 day level will be compared.
Beta-hydroxybutyrate | Baseline to 7 days
  Baseline to 7 day level will be compared.
Patient Reported Outcomes Measure Information System (PROMIS) - Physical Function | Baseline to 7 days
  This tool is a well-developed and validated method to obtain self-reported parameters of health in adults, we will be using: PROMIS® Item Bank v2.0 - Physical Function - Short Form 20a
  Subjects will rank 20 questions from a scale of 1 - 5, with 5 being the highest physical function and 1 being the lowest. The score will be added up, and the Raw score will be converted to T-Score using the PROMIS Adult v2.0 Physical Function 20a Short Form Conversion Table.
  Baseline to 7 day T-Score will be compared, with a Higher T-Score indicating higher physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Solis-Herrera, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected Individual Participant Data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At one year after study primary completion on ClinicalTrials.gov and at study completion at the time of publication in a peer review journal